CLINICAL TRIAL: NCT03486782
Title: Effect of Dual Site-dual Channel Non-invasive Brain Stimulation for Recovery of Language and Cognitive Function in Stroke Patients
Brief Title: Dual Site-dual Channel Non-invasive Brain Stimulation for Language and Cognitive Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-08-124-B
Record Dates: First submitted 2018-03-22; First posted 2018-04-03 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Aphasia; Cognitive Impairment
Keywords: transcranial direct current stimulation; dual stimulation
MeSH Terms: conditions — Stroke; Aphasia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual stimulation (Active Comparator): i) anodal stimulation of ipsilesional inferior frontal cortex and cathodal stimulation of contralesional supraorbital area ii) anodal stimulation on ipsilesional dorsolateral prefrontal cortex and cathodal stimulation of contralesional supraorbital area
  Interventions: Device: IFG stimulation; Device: DLPFC stimulation; Behavioral: aphasia therapy
- Single stimulation 1 (Active Comparator): i) anodal stimulation of ipsilesional inferior frontal cortex and cathodal stimulation of contralesional inferior frontal cortex
  Interventions: Device: IFG stimulation; Behavioral: aphasia therapy
- Single stimulation 2 (Active Comparator): i) anodal stimulation of ipsilesional inferior frontal cortex and cathodal stimulation of contralesional supraorbital area
  Interventions: Device: IFG stimulation; Behavioral: aphasia therapy

INTERVENTIONS:
Device: IFG stimulation — stimulating inferior frontal cortex with transcranial direct current stimulation for 30 minutes
Device: DLPFC stimulation — stimulating dorsolateral prefrontal cortex with transcranial direct current stimulation for 30 minutes
  Arms: Dual stimulation
Behavioral: aphasia therapy — aphasia therapy for 30 minutes during transcranial direct current stimulation

SUMMARY:
The aim of this study is to investigate the effect of dual site-dual channel non-invasive brain stimulation for recovery of language and cognitive function in post stroke patients. Simultaneous dual site-dual channel stimulation was applied by using two sets of transcranial direct current stimulation devices. All subjects will go through four conditions of transcranial direct current stimulation with for 30 minutes. Four conditions are 1) Dual stimulation: i) anodal stimulation on ipsilesional inferior frontal cortex, ii) anodal stimulation on ipsilesional dorsolateral prefrontal cortex. 2) Single stimulation 1: anodal stimulation on ipsilesional inferior frontal cortex and cathodal stimulation on contralesional inferior frontal cortex; 3) Single stimulation 2: anodal stimulation on ipsilesional inferior frontal cortex and cathodal stimulation on contralesional supraorbital area.

ELIGIBILITY:
Inclusion Criteria:

* left hemisphere involved stroke patients
* patients diagnoses as post stroke aphasia

Exclusion Criteria:

* history of psychiatric disease
* patients with metal implants
* history of epilepsy
* pregnancy
* skin defect at the site of electrode attachment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Changes in Korean Boston naming test | Baseline and after intervention (approximately 2 weeks)
  measures naming ability thorough picture naming test
Changes in Korean Western Aphasia Battery | Baseline and after intervention (approximately 2 weeks)
  assessment of language function and provide aphasia quotients

SECONDARY OUTCOMES:
Digit span test | Baseline and after intervention (approximately 2 weeks)
  measures memory span
Korea Montreal Cognitive Assessment | Baseline and after intervention (approximately 2 weeks)
  measure cognitive function
Korean Color Word Stroop test | Baseline and after intervention (approximately 2 weeks)
  measures selective attention and executive function
Controlled Oral Word Association Test | Baseline and after intervention (approximately 2 weeks)
  measure verbal fluency
Changes of Cortical activation | Baseline and after intervention (approximately 2 weeks)
  Cortical activation is measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany)
Changes in brain activation of resting-state and task functional MRI | Baseline and after intervention (approximately 2 weeks)
  Neuroplasticity measure

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided